CLINICAL TRIAL: NCT00005830
Title: Phase I Toxicity Trial of Doxorubicin-Cisplatin Followed by Whole Abdominal Irradiation for Advanced Endometrial Carcinoma
Brief Title: Combination Chemotherapy Plus Radiation Therapy in Treating Patients With Stage III or Stage IV Endometrial Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Gynecologic Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: GOG Foundation (Network)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GOG-9908; NCI-2012-02332 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000067844; GOG-9908 (Other: Gynecologic Oncology Group); GOG-9908 (Other: CTEP); U10CA027469 (NIH)
Record Dates: First submitted 2000-06-02; First posted 2003-01-27 (Estimated); Last update posted 2014-12-31 (Estimated); Status verified 2014-12

CONDITIONS: Endometrial Adenocarcinoma; Endometrial Clear Cell Adenocarcinoma; Endometrial Serous Adenocarcinoma; Stage III Uterine Corpus Cancer; Stage IV Uterine Corpus Cancer
MeSH Terms: interventions — Doxorubicin; Cisplatin; Radiotherapy; Radiation

ARMS (1):
- Treatment (doxorubicin, cisplatin, radiation therapy) (Experimental): Patients receive doxorubicin IV and cisplatin IV on day 1. Treatment repeats every 3 weeks for 3 courses. Patients then undergo whole abdominal radiotherapy 5 days a week for 4-6 weeks.
  Interventions: Drug: Doxorubicin Hydrochloride; Drug: Cisplatin; Radiation: Radiation Therapy

INTERVENTIONS:
Drug: Doxorubicin Hydrochloride — Given IV
Drug: Cisplatin — Given IV
Radiation: Radiation Therapy — Undergo radiation therapy
  Other Names: Cancer Radiotherapy; Irradiate; Irradiated; Irradiation; RT

SUMMARY:
Phase I trial to study the effectiveness of combination chemotherapy plus radiation therapy in treating women who have stage III or stage IV endometrial cancer. Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Radiation therapy uses high-energy x-rays to damage tumor cells. Combining chemotherapy with radiation therapy may kill more tumor cells.

DETAILED DESCRIPTION:
OBJECTIVES:

I. Determine the feasibility of doxorubicin and cisplatin followed by whole abdominal radiotherapy in patients with stage III or IV endometrial cancer.

II. Determine the acute and chronic toxic effects, in particular, severe and life-threatening gastrointestinal, hepatic, and hematologic toxic effects, of this regimen in these patients.

OUTLINE: This is a multicenter study.

Patients receive doxorubicin IV and cisplatin IV on day 1. Treatment repeats every 3 weeks for 3 courses. Patients then undergo whole abdominal radiotherapy 5 days a week for 4-6 weeks.

Patients are followed every 3 months for 2 years, every 6 months for 3 years, and then annually thereafter.

PROJECTED ACCRUAL: A total of 21-53 patients will be accrued for this study within 3.5 years.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed endometrial cancer including 1 of the following subtypes:

  * Clear cell carcinoma
  * Serous papillary carcinoma
  * Endometrioid adenocarcinoma
* Stage III or IV disease

  * Positive adnexa
  * Metastases to serosa, bowel mucosa, abdomen
  * Positive pelvic or paraaortic nodes
  * Positive pelvic washings or vaginal involvement within the radiation port
* Tumor must be surgically reduced to 2 cm or less within 8 weeks of study entry

  * Must have had a hysterectomy and bilateral salpingo oophorectomy
* No recurrent disease
* No distant metastases outside of abdominopelvic area, including:

  * Parenchymal liver metastases
  * Lung metastases
  * Positive inguinal lymph nodes
  * Positive supraclavicular nodes
  * Pleural effusion with malignant cytology
* Performance status - GOG 0-2
* Absolute neutrophil count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3
* Bilirubin no greater than 1.5 times upper limit of normal (ULN)
* SGOT and alkaline phosphatase no greater than 3 times ULN
* Creatinine no greater than ULN
* Cardiac ejection fraction greater than 50%
* No other prior or concurrent malignancy within the past 5 years except nonmelanoma skin cancer
* No prior chemotherapy
* No prior pelvic or abdominal radiotherapy
* No prior radiotherapy for other prior malignancy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2000-07; Primary Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
Number of patients completing the prescribed therapy | Up to 9 weeks
Frequency and severity of acute adverse effects as assessed by CTEP CTC version 2.0 | 3 weeks
Frequency and severity of chronic adverse effects as assessed by CTEP CTC version 2.0 | Up to 5 years after completion of study treatment
Frequency of severe and life threatening bowel, hepatic, and hematologic toxicity as assessed by CTEP CTC version 2.0 | Up to 9 weeks

SECONDARY OUTCOMES:
Reason for discontinuing study therapy | Up to 9 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Fowler, Principal Investigator — Gynecologic Oncology Group
Locations (1):
- Gynecologic Oncology Group, Philadelphia, Pennsylvania, United States